CLINICAL TRIAL: NCT07042906
Title: Comparison of the Factors Affecting PSI and BIS Values in Monitoring Anesthetic Depth During Open-Heart Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Mahsum Mazlum Mentes, residency doctor, Kocaeli University
Other Study IDs: GOKAEK-2023/06.13
Record Dates: First submitted 2025-05-14; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: BIS-EEG; PSI; Open Heart Surgery; Anesthesia Depth Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: anesthesia depth monitorizing, awareness — Investigation of BIS and PSI Monitoring Methods for Anesthetic Depth and the Factors Affecting These Methods in Open-Heart Surgery

SUMMARY:
Measurement of anesthetic depth has long been a subject of investigation, aiming to titrate anesthetic agents appropriately and to prevent intraoperative awareness and consciousness. Many patients undergoing surgery experience fear and anxiety regarding the possibility of remaining conscious, perceiving pain, and being unable to move during anesthesia. Intraoperative awareness-defined as consciousness during anesthesia with explicit recall afterward-is a distressing condition that can lead to post-traumatic stress disorder.

However, aiming for excessively deep anesthesia to avoid the possibility of awareness during surgery is not recommended, as it may result in hemodynamic instability due to the effects of anesthetic agents and may impair postoperative cognitive functions, particularly in the elderly population.

Common methods used in monitoring anesthetic depth include observing sweating, lacrimation, pupillary dilation, heart rate variability, and blood pressure. However, some of these are subjective and may not always be reliable indicators.

Electroencephalogram (EEG)-based monitors such as the Bispectral Index (BIS) and the Patient State Index (PSI) offer more reliable and objective means of monitoring anesthetic depth. These monitors provide numerical values between 0 (indicating unconsciousness) and 100 (indicating full alertness) based on proprietary algorithms, offering valuable insight into the patient's anesthetic state.

"Our aim is to examine BIS and PSI values and to investigate the factors that influence these parameters."

ELIGIBILITY:
Inclusion Criteria:

* "Patients aged 18 to 65 years,
* Classified as ASA (American Society of Anesthesiologists) physical status II-III,
* scheduled for elective open-heart surgery via median sternotomy

Exclusion Criteria:

* "Patients with an ejection fraction below 35%,
* Those with pre-existing central nervous system disorders (e.g., history of epileptic seizures or intracranial space-occupying lesions),
* A history of prior open cranial surgery,
* Known allergies to anesthetic agents, alcohol or substance abuse,
* Any other conditions deemed to negatively affect the BIS profile (e.g., patients with preoperative intra-aortic balloon pump insertion, those undergoing surgery under inotropic support, or receiving preoperative sedative infusions),
* As well as patients scheduled to undergo antegrade or retrograde cerebral perfusion or total circulatory arrest

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: "This study will be conducted with the approval of the Ethics Committee of Kocaeli University Faculty of Medicine Hospital and after obtaining written informed consent from all participants. The aim of our study is to investigate the factors influencing the BIS (Bispectral Index) and PSI (Patient State Index) methods, which are used to assess the depth of anesthesia in patients undergoing open-heart surgery with the use of a cardiopulmonary bypass (CPB) machine at Kocaeli University Faculty of Medicine Hospital."
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2025-07-18 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to measure the correlation between BIS and PSI values, which are parameters used to monitor the depth of anesthesia during open-heart surgery. | Data will be collected over a 12-month period and subjected to statistical analysis.
  BIS (Bispectral Index) is a monitoring method that uses EEG (electroencephalogram) data to measure the depth of anesthesia. It has been used for a long time to assess anesthetic depth. PSI (Patient State Index) is a monitoring method that has become more popular in recent years for measuring the depth of anesthesia. The recommended reference ranges for anesthetic depth are 40-60 for BIS and 25-50 for PSI. The primary objective of this study is to measure the correlation between PSI and BIS values during open-heart surgery.

SECONDARY OUTCOMES:
The secondary objective of this study is to measure the effect of hypothermia, which develops after patients are connected to the cardiopulmonary bypass (CPB) machine during open-heart surgery, on BIS and PSI values that indicate the depth of anesthesia | Data will be collected over a 12-month period and subjected to statistical analysis.
  BIS is a monitoring method that uses EEG (electroencephalogram) data to measure the depth of anesthesia. It has been used for a long time for this purpose. PSI is a monitoring method that has become more popular in recent years for assessing anesthetic depth. The recommended reference ranges for anesthetic depth are 40-60 for BIS and 25-50 for PSI. In the literature, there are studies suggesting that the decrease in body temperature (hypothermia) during cardiopulmonary bypass (CPB) in open-heart surgery is similar to the decrease observed in BIS and PSI values. In this study, our secondary objective is to measure the similarity between the decrease in body temperature and the decrease in BIS and PSI values.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Köseköy, Kocaeli, Turkey (Türkiye)